CLINICAL TRIAL: NCT04503733
Title: A Randomized, Double-blind, Placebo-Controlled, Dose Escalation Study to Assess Safety, Efficacy and Pharmacokinetics of GMA301 in Subjects With Pulmonary Arterial Hypertension
Brief Title: A Study of GMA301 in Subjects With Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gmax Biopharm LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GETA_MAD_01
Record Dates: First submitted 2020-07-24; First posted 2020-08-07 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Q4W GMA301 IV injections (300 mg) (Experimental): Drug: Q4W GMA301 IV injections (300 mg) Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Other: Q4W placebo IV injections Placebo is indistinguishable from GMA301
  Interventions: Drug: Q4W GMA301 IV injections (300 mg); Other: Q4W placebo IV injections
- Q4W GMA301 IV injections (600 mg) (Experimental): Drug: Q4W GMA301 IV injections (600 mg) Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Other: Q4W placebo IV injections Placebo is indistinguishable from GMA301
  Interventions: Drug: Q4W GMA301 IV injections (600 mg); Other: Q4W placebo IV injections
- Q4W GMA301 IV injections (1000 mg) (Experimental): Drug: Q4W GMA301 IV injections (1000 mg) Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Other: Q4W placebo IV injections Placebo is indistinguishable from GMA301
  Interventions: Drug: Q4W GMA301 IV injections (1000 mg); Other: Q4W placebo IV injections
- Q4W GMA301 IV injections (1800 mg) (Experimental): Drug: Q4W GMA301 IV injections (1800 mg) Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Other: Q4W placebo IV injections Placebo is indistinguishable from GMA301
  Interventions: Drug: Q4W GMA301 IV injections (1800 mg); Other: Q4W placebo IV injections

INTERVENTIONS:
Drug: Q4W GMA301 IV injections (300 mg) — Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Arms: Q4W GMA301 IV injections (300 mg)
Drug: Q4W GMA301 IV injections (600 mg) — Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Arms: Q4W GMA301 IV injections (600 mg)
Drug: Q4W GMA301 IV injections (1000 mg) — Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Arms: Q4W GMA301 IV injections (1000 mg)
Drug: Q4W GMA301 IV injections (1800 mg) — Each cohort will contain 12 subjects, 9 of whom will be administered active GMA301 and 3 of whom will be administrated placebo.
  Arms: Q4W GMA301 IV injections (1800 mg)
Other: Q4W placebo IV injections — Placebo is indistinguishable from GMA301.

SUMMARY:
A Randomized, Placebo-Controlled, Double-blind, Dose Escalation Study to Assess Safety, Efficacy and Pharmacokinetics of GMA301 Injection in Subjects with Pulmonary Arterial Hypertension

DETAILED DESCRIPTION:
Drug: Q4W GMA301 IV injections (300 mg) Drug: Q4W GMA301 IV injections (600 mg) Drug: Q4W GMA301 IV injections (1000 mg) Drug: Q4W GMA301 IV injections (1800 mg) Other: Q4W placebo IV injections

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Male or female, aged 18 to 75 years inclusive
2. WHO Group 1 PAH related to one of the following conditions:

   1. Idiopathic
   2. Heritable
   3. Drugs or toxins-induced
   4. Associated with connective tissue disease
   5. Associated with congenital heart disease if subjects underwent surgical correction more than 12 months before Screening
3. Symptoms due to PAH are consistent with WHO functional class II- III
4. Have not taken endothelin receptor antagonists (ERAs) within 3 months before Randomization
5. Has been taking at least one oral PAH targeted drug that has been approved by local guidelines for at least 3 months before Screening with stable dosage and the disease did not worsen during this period per Investigator's judgment
6. Right heart catheterization (RHC) result meets below criteria when Screening:

   1. Mean pulmonary arterial pressure (PAP) ≥25 mmHg
   2. Pulmonary vascular resistance (PVR) >3 Woods units
   3. PA wedge pressure (PAWP) ≤15 mmHg

   If a subject has undergone RHC within 3 months before Screening, the waveform results will serve as baseline data only if they meet the entry criteria and the RHC at Screening will not be repeated. In case PAWP cannot be well measured during RHC, left ventricular end diastolic pressure will be tested by left heart catheterization.
7. Has a six-minute walk test (6MWT) with distance between 150 to 450 meters at Screening
8. The dosage of digitalis drugs or L-arginine supplementation must be stable for at least 1 month before Screening, if applicable.
9. No new use of an IV diuretic, cardiotonic (positive inotropic agents), or vasoactive drug within 30 days before Screening
10. Both male and female subjects agree to use 2 medically acceptable methods of contraception (Appendix 4) throughout the entire study period from informed consent signing to 90 days after last dose, if the possibility of conception exists. Medically acceptable methods of contraception include oral, implantable, or injectable contraceptives (starting 2 months before dosing); diaphragm with vaginal spermicide; intrauterine device; condom and partner using vaginal spermicide; and surgical sterilization (6 months after surgery). Women who are surgically sterile or those who are postmenopausal for at least 2 years are not considered to be of childbearing potential. Eligible male and female subjects must agree not to participate in a conception process (i.e. active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) during the study and for 90 days after the last dose of study drug.
11. Body weight no less than 40 kg at Screening
12. Able to understand and willing to sign the Informed Consent Form (ICF) and comply with the study procedures.

Exclusion Criteria

Subjects who me et any of the following criteria will not be allowed to participate in this study:

1. Diagnosed with WHO Group II, III, IV, V of PH
2. Use of calcium channel blockers within 1 month prior to Screening
3. Systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg at Screening
4. SBP <90 mmHg at Screening
5. Pulmonary function test: FEV1 <60% of predicted, TLC <60% of predicted, DLCO <60% of predicted
6. History of pulmonary embolism as judged by the Investigator
7. Uncontrolled sleep apnea at the discretion of the Investigator
8. Limited full participation in the 6MWT due to arthritic, neuromuscular, vascular or other diseases unrelated to PAH
9. History of acute cardiovascular and/or cerebrovascular events within 6 months before Screening
10. Echocardiogram (ECHO) demonstrating at least one of the following at Screening:

    1. LVEF <50%
    2. Mean end-diastolic left ventricular septal and posterior wall thickness of >12 mm
    3. Left atrial (LA) area on apical 4 chamber view >20 cm2
    4. LA volume >55 mL
    5. LA volume index >34 mL/m2
    6. Significant valvular heart disease including moderate or severe mitral or aortic stenosis with an aortic valve area <1.0 cm2 or mitral valve area <1.5 cm2, greater than moderate aortic or mitral regurgitation, greater than moderate tricuspid or pulmonic stenosis
11. Restrictive, dilated or hypertrophic cardiomyopathy or constrictive pericarditis
12. Using non-oral prostacyclin when Screening
13. Laboratory parameters during Screening:

    1. Baseline aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 times the upper limit of normal (ULN) or total bilirubin ≥1.5 times ULN
    2. Estimated glomerular filtration rate (eGFR) <60 mL/min by Cockcroft-Gault formula

       Online calculation available from https://www.kidney.org/professionals/KDOQI/gfr_calculatorCoc

       Cockcroft-Gault formula (1973):

       Male: CCr=((l40-Age) × Weight)/(72×SCr)

       Female: CCr={((l40-Age) × Weight)/(72×SCr)}× 0.85

       CCr (creatinine clearance rate) = mL/min

       Age = year

       Weight = Kg

       SCr (serum creatinine) = mg/dL
    3. Hemoglobin concentration ≤100 g/L at Screening
14. QTc interval by Fridericia's criteria (QTcF) ≥500 msec at Screening
15. Malignancy within 5 years before Screening visit (with the exception of localized non-metastatic basal cell carcinoma of the skin, non-metastatic carcinoma of the prostate or in-situ carcinoma of the cervix excised with curative results)
16. Alcohol or drug abuse within 1 year before Screening
17. A psychiatric, addictive or other disorder that compromises the ability to give informed consent for participating in this study
18. History of organ transplantation
19. Pregnant or nursing females
20. History of HIV
21. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or HIV antibody (HIV-ab)
22. Enrolled in another interventional study within 30 days before Screening
23. Any condition that, in the opinion of the Investigator, prevents a potential subject from safely participating in the study
24. Start a new exercise program or participate in any unusually strenuous physical exertion within 6 weeks prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-10-26 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of Treatment-emergent Adverse Events (TEAE) in subjects assigned to GMA301 compared with those assigned to placebo. | Through study completion (up to 22 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics (Area under the serum concentration- time curve from time zero to the last measurable concentration) | Through study completion (up to 22 weeks)
Comparison of GMA301 treatment effect at Week 12 versus baseline regarding the pulmonary vascular resistance (PVR) based on right heart catheterization (RHC) | Baseline to Week 12
Comparing 6MWT distance | Baseline to Week 12

OTHER OUTCOMES:
Changes in REVEAL 2.0 risk score at Week 12 compared with baseline | Baseline to Week 12
  Calculated risk scores can range from 0 (lowest risk) to 23 (highest risk).

CONTACTS AND LOCATIONS:
Overall Officials: Hua Yao, Principal Investigator — Guangdong Provincial People's Hospital; Lan Wang, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Wei Huang, Principal Investigator — First Affiliated Hospital of Chongqing Medical University; Zaixin Yu, Principal Investigator — Xiangya Hospital of Central South University; Fenling Fan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Zhicheng Jing, Principal Investigator — Peking Union Medical College Hospital - Dongcheng District; Aaron Waxman, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- China (6):
  - Peking Union Medical College Hospital - Dongcheng District, Beijing
  - Xiangya Hospital, Central South University, Changsha
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangdong General Hospital, Guangzhou
  - Shanghai Pulmonary Hospital, Shanghai
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04503733/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04503733/ICF_001.pdf